CLINICAL TRIAL: NCT00003321
Title: An International Field Study of the Reliability and Validity of the EORTC-QLQ-C30 and a Disease Specific Questionnaire Module (the EORTC OES-24) in Assessing the Quality of Life of Patients With Oesophageal Cancer
Brief Title: Quality-of-Life Assessment of Patients Who Have Cancer of the Esophagus
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-15961-40973; EORTC-15961/40973
Record Dates: First submitted 1999-11-01; First posted 2004-03-22 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Esophageal Cancer
Keywords: stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Questionnaires that measure quality of life may improve the ability to plan treatment for patients who have cancer of the esophagus.

PURPOSE: This clinical trial studies quality-of-life assessments of patients with cancer of the esophagus who are receiving treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Test the psychometric, clinical, and cross cultural validity and reliability of the quality-of-life questionnaire EORTC-QLQ-C30 (version 3.0) in conjunction with the esophageal cancer-specific module EORTC QLQ-OES-24 in patients with esophageal cancer.

OUTLINE: This is a multicenter study. Patients are stratified by treatment (potentially curative vs purely palliative). Patients receiving potentially curative treatment are further stratified according to study treatment (esophagectomy alone vs esophagectomy plus adjuvant or neoadjuvant chemo/radiotherapy vs radical radiotherapy with or without chemotherapy). Patients receiving purely palliative treatment are further stratified according to study treatment (intubation/laser/ethanol injection vs palliative chemo/radiotherapy without endoscopic relief of dysphagia). Patients are administered two questionnaires: (1) The EORTC QLQ-C30 (version 3.0) is a 30-item questionnaire about patient ability to function, symptoms related to the cancer and its treatment, overall health and quality of life, and perceived financial impact of the cancer and its treatment. (2) The EORTC QLQ-OES-24 is a 24-item esophageal cancer-specific questionnaire supplementing EORTC QLQ-C30 with information about disease and treatment-related symptoms and side effects, dysphagia, nutrition, and social and emotional effects of esophageal cancer. Both questionnaires are administered once before and once during or after treatment.

PROJECTED ACCRUAL: 370 patients (170 with locoregional disease, 200 with metastatic disease) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Group I: Local or locoregional primary esophageal or esophago-gastric cancer Planned esophagectomy with or without adjuvant or neoadjuvant chemotherapy and/or radiotherapy OR Planned radical radiotherapy with or without chemotherapy Prior endoscopic procedure to relieve dysphagia allowed No distant liver or bone metastasis if undergoing esophagectomy Group II: Metastatic esophageal cancer or local anastomotic recurrence of esophageal cancer or deemed unsuitable for esophagectomy Prior palliation by endoscopic or open intubation, laser treatment, tumor necrosis with alcohol injection or diathermy, or intraluminal radiotherapy allowed Prior palliative radiotherapy or chemotherapy allowed No cerebral metastases

PATIENT CHARACTERISTICS: Age: Any age Performance status: Not specified Life expectancy: Group I: At least 3 months Group II: At least 4 weeks Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Mentally fit to complete a questionnaire or undergo an interview Aware of diagnosis No concurrent second malignancy except basal cell skin cancer No concurrent participation in other quality-of-life studies

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 1998-02; Primary Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Blazeby, MB, CHB, FRCS, BSc, MD, Study Chair — University Hospitals Bristol and Weston NHS Foundation Trust
Locations (10):
- Sir Charles Gairdner Hospital, Perth, Perth, Western Australia, Australia
- France (2):
  - Clinique Armoricaine De Radiologie, Saint Brieux
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (2):
  - Robert Roessle Klinik, Berlin
  - University of Marburg, Marburg
- Diakonissehjemm Ets University Hospital, Bergen, Norway
- Hospital De Navarra, Pamplona, Spain
- Sahlgrenska University Hospital, Gothenburg (Goteborg), Sweden
- Hopital Cantonal Universitaire de Geneva, Geneva, Switzerland
- Bristol Royal Infirmary, Bristol, England, United Kingdom

REFERENCES:
- [Background] Conroy T, Etienne PL, Adenis A, Ducreux M, Paillot B, Oliveira J, Seitz JF, Francois E, Van Cutsem E, Wagener DJ, Kohser F, Daamen S, Praet M, Gorlia T, Baron B, Wils J; European Organisation for Research and Treatment of Cancer Gastrointestinal Tract Cancer Cooperative Group. Vinorelbine and cisplatin in metastatic squamous cell carcinoma of the oesophagus: response, toxicity, quality of life and survival. Ann Oncol. 2002 May;13(5):721-9. doi: 10.1093/annonc/mdf063. PMID 12075740